CLINICAL TRIAL: NCT05279261
Title: Clinical Effect of the Axillary Approach to Acute Anterior Glenoid Fractures
Brief Title: Clinical Effect of the Axillary Approach to Glenoid Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00006761-M2019363
Record Dates: First submitted 2021-07-01; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2021-07

CONDITIONS: Fracture; Glenoid
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Undergo the axillary approach
  Interventions: Procedure: The axillary approach

INTERVENTIONS:
Procedure: The axillary approach — The approach enters from the axilla through the interval between the latissimus dorsi and subscapularis to expose the anteroinferior glenoid, neck and lateral border of the scapula with entire rotator cuff sparing and fix the fracture with screws or plates.

SUMMARY:
Glenoid fractures result in glenohumeral post-trauma arthritis and instability. Operative treatment is indicated for severe fractures. The traditional deltopectoral approach, which requires detachment of the subscapularis, has many drawbacks, including loss of external rotation and suboptimal fixation. Arthroscopic techniques also cannot allow anatomic reduction and biomechanical stability for large fractures. We describe an alternative approach that enters from the axilla through the interval between the rotator cuff and the inferior glenoid, neck and lateral border of the scapula without detachment of the rotator cuff.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic and closed fractures
* Fracture type conforms to Ideberg Ia classification or AO/OTA F1.1 classification
* Fracture displacement ≥4mm, the area of involvement ≥20%.

Exclusion Criteria:

* Severe multiple trauma
* Pathological fracture
* Unable to tolerate surgical treatment
* The interval between injury and operation was > 2 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-06-12 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
fracture union | 6 months
  X-rays and CT scans are used to evaluate the bone union
the Constant and Murley scores | 2 years
  The questionaire evaluates shoulder function in terms of pain (15 points), daily activities (20 points), range of motion (40 points) and muscle strength (25 points) on a scale of 100, with the higher the score, the better the function.
the DASH(disabilities of the arm，shoulder and hand) scores | 2 years
  Shoulder function was evaluated by patients' subjective feelings about pain, activity, daily life, work and entertainment of the affected limb in the past 1 week. A total of 30 items were evaluated, and the score of each item was 1-5, DASH= (total score-30) /1.2, with the maximum score of 100, the lower the score, the better the function

SECONDARY OUTCOMES:
Complications | 2 years
  The presence of postoperative complications,including implant failure, osteolysis, and soft-tissue reactions, are determined by symptoms and images.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospita, Beijing, China